CLINICAL TRIAL: NCT04876482
Title: Efficacy of Oropharyngeal Myofunctional Therapeutic Training for Obstructive Sleep Apnea Patients After Transoral Robotic Surgery
Brief Title: Myofunctional Training for Obstructive Sleep Apnea Patients After Transoral Robotic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKUH-10902002
Record Dates: First submitted 2021-02-03; First posted 2021-05-06 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2021-09

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Without the willingness of surgery, those participants waiting for oral appliance (Device), losing weights and using continuous positive airway pressure (Device) were distribute to control group.
  Interventions: Device: oral appliance; Device: using continuous positive airway pressure; Behavioral: losing weights
- Transoral robotic surgery (TORS) (Experimental): The participants underwent TORS. TORS is a kind of surgery that the surgeons would remove the tonsils and the fat tissue of tongue base and suspend the soft palate.
  Interventions: Procedure: transoral robotic surgery
- TORS+OPR (Experimental): The participants started OPR 6 weeks after TORS. Each exercise was repeated 10 times, 1-3 cycles per day, 3-5 sessions per week at their home and performed for 3 months. Patients were supervised by physical therapist once a week for 30 minutes.
  Interventions: Procedure: transoral robotic surgery; Combination Product: oropharyngeal rehabilitation

INTERVENTIONS:
Procedure: transoral robotic surgery — transoral robotic surgery (TORS) which remove the extra soft tissue of the base of the tongue and soft palate in this study
  Arms: TORS+OPR; Transoral robotic surgery (TORS)
Device: oral appliance — It is a kind of treatment for the participants who refuse surgeries and choose to use other kinds of conservative treatment. The conservative treatments included oral appliance, losing weights and using continuous positive airway pressure. The oral appliance would be wore only at night and it would press the soft palate and protrude the jaw.
  Arms: Control
Device: using continuous positive airway pressure — The participants only used CPAP at night. The device composed of a main machine, pipe and mask. The participants would instruct to wore the mask. The main machine would give positive airway pressure to open the airway and avoid collapsing.
  Other Names: CPAP
  Arms: Control
Behavioral: losing weights — The participants would ask to lose weight by changing their diets and exercising, without using drugs and surgeries.
  Arms: Control
Combination Product: oropharyngeal rehabilitation — OPR included exercise for soft palate, tongue and oropharynx. There are 13 movements in OPR. The movements would be teach by a physical therapist.
  Other Names: OPR
  Arms: TORS+OPR

SUMMARY:
Background: Obstructive Sleep Apnea Syndrome (OSA) is a kind of sleep disorder. The symptoms are intermittent, partial or complete upper airway collapse, seriously impacting oxygen saturation and oxidative stress. Some patients choose to do upper airway surgeries, but the success rate is only 60-70%. The symptoms might relapse because of aging and gaining weights. The purpose of our study is to compare the effect of transoral robotic surgery (TORS) and oropharyngeal rehabilitation (OPR) on patients after TORS. Methods: Participants above 20 years old who are newly diagnosed with mild to severe OSA (Apnea-hypopnea Index >5/h), and the physician will explain the treatment programs to every subject in clinic. Expected results: The hypothesis of this study is the success rate of surgery will be enhance by increasing tongue and jaw-opening muscle strength after OPR. The biomarkers of cardiovascular disease may decrease and both the collapse of upper airway and sleep quality may be improved after TORS and OPR.

DETAILED DESCRIPTION:
The participants above 20 years old who are newly diagnosed with mild to severe OSA (Apnea-hypopnea Index >5/h), and the physician will explain the treatment programs to every subject. By their willingness to choose the therapeutic method, the participants who select the surgery interventions will be assign to TORS or TORS+OPR group. The matched controls as well as age-, sex-, and body mass index-matched OSA participants will be selected from the patients who are waiting for oral appliance, losing weight and using continuous positive airway pressure. Before surgery, 6 week and 18 week after surgery, the investiagters will compare the polysomnography data, questionnaires of sleep quality, drug-induced sleep endoscopy and computed tomography as primary outcomes. The investigators will also compare the tongue and jaw-opening muscle strength and biomarkers of oxidative stress, anti-oxidative stress, inflammatory cytokines and matrix metalloproteinases 9 as secondary outcomes. The OPR would begin at 6 week after surgery, and participants will undergo three months of the home-based oropharyngeal myofunctional therapeutic training. During the training intervention period, participants will be interviewed one time per week for adjusting the treatment intensity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to severe OSA in the past year
* Age between 20-65 years old.

Exclusion Criteria:

* A history of malignancy or infection of the head and neck region and laryngeal trauma
* Craniofacial malformation
* Stroke
* Neuromuscular disease
* Heart failure
* Coronary artery disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited time:2020/01/01-2022/05/11
Period: Overall Study
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Started | 20 | 42 | 19
Completed | 17 | 38 | 19
Not Completed | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR | Total
Number analyzed (Participants) | 20 | 42 | 19 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 42 | 19 | 81
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.25 (9.55) | 43.12 (10.87) | 45.10 (8.63) | 43.91 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 11
  Male | 15 | 37 | 18 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 42 | 19 | 81
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 20 | 42 | 19 | 81
Polysomonography [Mean (Standard Deviation); unit: events per hour] — Apnea hypopnea index (AHI) is the main measurement, so the mean and SD below was for AHI.
  Apnea was defined as a reduction in airflow >90% lasting >10 seconds.The definition of hypopnea was a reduction in airflow >30% lasting >10 seconds and a decrease in oxygen saturation >3% or presence of microarousal. AHI quantifies the severity of sleep apnea by counting the number of apneas and hypopneas during sleep. Mild sleep apnea means 5< =AHI<15; Moderate sleep apnea means 15< =AHI<30; Severe sleep apnea means AHI >=30
  events per hour | 38.39 (22.15) | 43.98 (19.86) | 45.43 (21.71) | 42.92 (20.86)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — using weight and height and the formula is kg/m^2
  kg/m^2 | 27.11 (3.48) | 28.09 (3.72) | 27.31 (4.18) | 27.62 (3.76)
Neck circumference [Mean (Standard Deviation); unit: cm] — Using the unit as centimeter
  cm | 37.81 (2.53) | 39.38 (3.48) | 39.53 (2.08) | 39.00 (2.98)
Tongue protrusion muscle strength [Mean (Standard Deviation); unit: kPa] | 52.50 (12.82) | 61.16 (16.94) | 51.00 (15.87) | 56.10 (16.17)
Tongue elevation muscle strength [Mean (Standard Deviation); unit: kPa] | 52.50 (14.13) | 58.25 (15.25) | 50.47 (10.52) | 54.61 (14.05)
Tongue depression muscle strength [Mean (Standard Deviation); unit: kPa] | 43.56 (10.19) | 47.16 (11.04) | 40.95 (10.86) | 44.51 (10.95)
Tongue lateralization muscle strength [Mean (Standard Deviation); unit: kPa] | 35.72 (9.98) | 42.20 (11.81) | 41.79 (11.45) | 40.40 (11.44)
Computed Tomography_ Volume [Mean (Standard Deviation); unit: cm^3] — Volume from hard palate to epiglottis tip
  cm^3 | 19.04 (11.40) | 19.33 (8.67) | 16.80 (6.07) | 18.56 (8.82)
Computed Tomography_ minimal area [Mean (Standard Deviation); unit: cm^2] — Minimal area on the epiglottis tip
  cm^2 | 3.71 (1.94) | 3.88 (1.44) | 3.54 (1.38) | 3.74 (1.55)
Computed Tomography_ AP distance [Mean (Standard Deviation); unit: cm] — Anterior to posterior distance on epiglottis tip
  cm | 1.72 (0.77) | 1.70 (0.49) | 1.66 (0.40) | 1.69 (0.55)
Computed Tomography_ lateral distance distance [Mean (Standard Deviation); unit: cm] — Left to right distance on epiglottis tip. Unit was measured in centimeter.
  cm | 3.02 (0.84) | 3.30 (0.74) | 3.22 (0.51) | 3.20 (0.71)
Drug-induced sleep endoscopy [Count of Participants; unit: Participants] | 20 | 42 | 19 | 81
Jaw opening muscle strength [Mean (Standard Deviation); unit: kg] | 8.97 (3.70) | 9.70 (3.87) | 9.84 (2.52) | 9.55 (3.47)

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: Polysomnography included electroencephalographic, electro-oculographic, thoracic and abdominal respiratory inductance plethysmography and body position sensor to confirm the sleeping stage in one-night observation. Above measurements will be aggregated to arrive AHI.
  Unabbreviated scale title:Apnea and Hypopnea index The minimum value:0 The maximum values: none Higher scores mean a worse outcome.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
events per hour | 44.89 (21.09) | 44.65 (19.91) | 36.87 (21.87)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the AHI would be higher in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — The Overall Number of Participants Analyzed do not appear to be equal, so we used linear regrssion to compare the mean difference among three groups; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -10.76

2. Primary Outcome: Computer Tomography (CT)_Volume
Description: All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Volume from hard palate to the base of epiglottis was measured.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
cm^3 | 18.39 (11.47) | 18.72 (6.43) | 16.80 (6.07)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the upper airway volume would be higher in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 2.05

3. Primary Outcome: Computer Tomography (CT)_minimal Area
Description: All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Cross section area on the tip of epiglottis was measured.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 42 | 19
cm^2 | 3.60 (1.94) | 3.80 (1.13) | 3.54 (1.38)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the minimal area on the tip of epiglottis would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.275

4. Primary Outcome: Computer Tomography (CT)_AP Distance
Description: All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Anterior to posterior distance on the tip of epiglottis was measured.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
cm | 1.71 (0.79) | 1.64 (0.39) | 1.66 (0.40)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the anteror to posterior distance on the tip of epiglottis would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -0.14

5. Primary Outcome: Computer Tomography (CT)_Lateral Distance
Description: All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Lateral distance on the tip of epiglottis was measured.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
cm | 2.92 (0.83) | 3.43 (0.63) | 3.22 (0.51)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the lateral distance on the tip of epiglottis would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.01

6. Primary Outcome: Drug-induced Sleep Endoscopy (DISE)
Description: All patients underwent DISE in a supine position. The possible outcomes were unilevel collapse at the velum, oropharynx, tongue base, or epiglottis and multilevel collapse at any of these locations. The velum is the part of the upper airway at the level of the soft palate and uvula; the oropharynx is the pharyngeal portion at the level of the tonsils, above the tongue base. The tongue base was considered the retroglossal area; epiglottis was considered the pharyngeal region below the tongue base. The degree of obstruciton was diagnosed by an ear nose throat surgeon. The degree of obstruction ranged from 0 to 2. 0: no obstruction (<50%); 1: partial obstruction (50-75%); 2: complete obstruction (>75%).
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
Participants
  The degree of obstruction in velum: no obstruction | 0 | 0 | 1
  The degree of obstruction in velum: partial obstruction | 9 | 6 | 7
  The degree of obstruction in velum: complete obstruction | 8 | 32 | 11
  The degree of obstruction in oropharynx: no obstruction | 2 | 2 | 1
  The degree of obstruction in oropharynx: partial obstruction | 13 | 28 | 13
  The degree of obstruction in oropharynx: complete obstruction | 2 | 8 | 5
  The degree of obstruction in tongue base: no obstruction | 0 | 0 | 1
  The degree of obstruction in tongue base: partial obstruction | 7 | 16 | 9
  The degree of obstruction in tongue base: complete obstruction | 10 | 22 | 9
  The degree of obstruction in epiglottis: no obstruction | 0 | 0 | 0
  The degree of obstruction in epiglottis: partial obstruction | 6 | 18 | 11
  The degree of obstruction in epiglottis: complete obstruction | 11 | 20 | 8
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that TORS followed by OPR would improve upper airway obstruction more compared with TORS alone and conservative treatment (control); Test type: Other — Baseline characteristics among the study groups were compared using Fisher exact test for categorical variables. McNemar chi-square test used for within-group analysis; p < 0.05, Fisher Exact; Number and percentage = 0.05

7. Primary Outcome: Jaw Opening Muscle Strength
Description: Muscle strength of jaw was measured with a 'handheld' dynamometer (MicroFET○R2, Hoggan Scientific, USA) mounted on an adapted ophthalmic examination frame, to avoid alterations in chin and head position and to ensure consistent compression.
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: kilogram force
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
kilogram force | 9.14 (3.67) | 9.63 (3.59) | 9.68 (2.49)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the jaw opening muscle strength would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 2.23

8. Primary Outcome: Tongue Protrusion Muscle Strength
Description: The muscle strength of the tongue was evaluated by the IOPI system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA).
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
kilopascals | 57.83 (11.17) | 56.97 (11.72) | 61.89 (8.88)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the tongue protrusion muscle strength would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 2.45

9. Primary Outcome: Tongue Elevation Muscle Strength
Description: The muscle strength of the tongue was evaluated by the IOPI system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA).
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
kilopascals | 59.17 (13.64) | 57.22 (12.59) | 63.37 (12.07)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the tongue elevation muscle strength would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 4.81

10. Primary Outcome: Tongue Depression Muscle Strength
Description: The muscle strength of the tongue was evaluated by the IOPI system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA).
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
kilopascals | 49.94 (10.22) | 48.22 (10.38) | 58.58 (9.16)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the tongue depression muscle strength would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 7.01

11. Primary Outcome: Tongue Lateralization Muscle Strength
Description: The muscle strength of the tongue was evaluated by the IOPI system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA).
Time Frame: through study completion, an average of 6 months
Population: Seven participants didn't complete the whole protocol, so we didn't analyze their data.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
Number analyzed (Participants) | 17 | 38 | 19
kilopascals | 42.19 (10.52) | 41.55 (9.86) | 50.11 (9.38)
Statistical Analysis 1: Comparison: Control vs Transoral Robotic Surgery (TORS) vs TORS+OPR; We hypothesized that the improvements in the tongue lateralization muscle strength would be more in patients who underwent TORS combined with OPR than in those who underwent only TORS and those who received conservative treatment (controls); Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 3.67

ADVERSE EVENTS:
Time Frame: 6 months
Description: None of the participants at risk for serious adverse events and all-cause mortality is zero becaurse control group only used conservative treatment and TORS is a safe surgery for surgery group and surgery + OPR group.
Arm/Group | Control | Transoral Robotic Surgery (TORS) | TORS+OPR
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/42 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/42 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/42 | 0/19

LIMITATIONS AND CAVEATS:
1. The small sample size of 78 participants with OSA, a higher number of male participants, and the inclusion of only participants of Asian ethnicity
2. Including patients who appeared motivated to undergo OPR in Group SO was likely to exaggerate the effectiveness of OPR because the patients might increase the frequency of OPR
3. Participant compliance in home-based exercise was monitored mainly through self-report
4. The intervention period of our OPR protocol was only 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04876482/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT04876482/ICF_001.pdf